CLINICAL TRIAL: NCT07118592
Title: Genetic Architecture of Natriuretic Peptides and Blood Pressure Response
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Associate Professor, Division of Cardiovascular, Department of Medicine, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300015234
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hypertension (HTN); Cardiometabolic Diseases
Keywords: Hypertension; Natriuretic peptides; Polygenic risk score; Cardiometabolic diseases
MeSH Terms: conditions — Hypertension; Genetic Risk Score | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Natriuretic Peptide Polygenic Score (Experimental): Active Comparator: High NP PGS Group
  Interventions: Dietary Supplement: Low Salt Diet; Dietary Supplement: High Salt Diet; Dietary Supplement: Saline Infusion
- Low Natriuretic Peptide Polygenic Score (Experimental): Experimental: Low NP PGS Group
  Interventions: Dietary Supplement: Low Salt Diet; Dietary Supplement: High Salt Diet; Dietary Supplement: Saline Infusion

INTERVENTIONS:
Dietary Supplement: Low Salt Diet — 8 days of diet with low salt content will be given to the study participants
Dietary Supplement: High Salt Diet — 8 days of diet with high salt content will be given to the study participants
Dietary Supplement: Saline Infusion — 2 Liters of normal saline infusion (0.25 ml/kg/min over 2 hours) will be given to the study participants at the end of each study period

SUMMARY:
Natriuretic peptides (NPs) are hormones produced by the heart and play an important role in maintaining cardiovascular health and have favorable metabolic benefits. Low NP levels are associated with an increased likelihood of the development of cardiometabolic diseases like diabetes and hypertension. NP levels are known to be highly heritable, with up to half of the differences in NP levels being explained by genetics. The investigators aim to describe the genetic architecture of NPs by examining the genetic variants associated with NPs, and generate and validate a polygenic score (PGS) for NPs. The investigators will use this NP PGS to examine the association of genetically determined NP levels with cardiometabolic and cardiovascular outcomes. The investigators will conduct a genotype-guided physiological clinical trial that aims to assess the genetic factors affecting NP levels and their impact on blood pressure and NP response to saline infusion, high-salt diet, and low-salt diet. These findings will help support personal medicine approaches to lower the increasing burden of hypertension in the United States.

DETAILED DESCRIPTION:
NPs are vital cardiac-derived hormones that are known for their role in salt regulation, vascular function, and blood pressure (BP) regulation. NPs are also key regulators of insulin sensitivity, lipid metabolism, and energy expenditure. Recent evidence has shown that low NP levels are associated with higher risk of cardiometabolic diseases like hypertension (HTN). Animal studies have shown that the loss of the NP gene in mice is associated with the development of salt-sensitive HTN. Prior research indicates that individuals with genetically lower NP levels show higher systolic and diastolic BP and are at a 15% higher risk of HTN.

NP levels are highly heritable, with heritability ranging from 35%-44%, independent of factors like age, body mass index, sex, and race. The availability of whole genome sequencing (WGS) data from a comprehensive cohort of individuals provides an opportunity to advance the discovery of novel genomic loci and rare variants regulating NP levels. Previous studies on the genetic determinants of NP levels were limited by their focus on diseased populations, use of genotyping array data, or lack of comprehensive genetic analysis. Examination of the genotype-based differences in NP may provide not only insights into the pathophysiology of diseases like salt-sensitive HTN, but also help discover new pharmacogenomic treatment approaches.

In the proposed study, the investigators will leverage data from multiple large cohorts, including the TransOmics for Precision Medicine cohorts, UK Biobank, and All of Us Research Program, to investigate the genetic architecture of NP levels, including the common, rare, and structural variants. The investigators will conduct fine mapping to identify variants that might cause disease and perform analyses to prioritize genes associated with NPs. Additionally, the summary statistics of the common variant analysis will be used to develop NP polygenic risk scores using standardized methodologies. The best-performing NP PGS will be validated, and the association of genetically determined NP levels with cardiometabolic and cardiovascular disease will be examined. The NP PGS will then be used to conduct a Mendelian randomization analysis to examine the causal role of NPs in cardiometabolic disease.

The investigators will enroll 200 hypertensive participants for 4 weeks, during which the participants will receive 1 week each of high and low-salt diets in a random sequence, and undergo a volume loading using a normal saline infusion protocol at the end of each diet period. Each diet period will be followed by a week of washout.

The investigators hypothesize that individuals with genetically determined low NP levels will exhibit a poorer response to salt and volume loading. The main questions this study aims to answer are:

* How does the genetic makeup of NP affect the BP differences after consuming a high and low salt diet?
* How do the NP precursor levels change following consumption of a high and low salt diet in participants with differences in genetically determined NP levels?

Using this NP PGS, the investigators will explore the clinical implications of genetically determined NP levels on the BP response to salt and volume loading by conducting a genotype-first trial, and this data will provide an understanding of the determinants of BP response and may foster new NP based individualized therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 18 years
* Consenting to collection of genetic material and willing to adhere to study protocol
* Stage I/II Hypertension (Systolic blood pressure: 130-159 and Diastolic blood pressure: 80-99 mm Hg)

Exclusion Criteria:

* Body mass index (BMI) more than 45 kg/m2
* History of uncontrolled hypertension (i.e., Systolic blood pressure more than or equal to 160 mmHg and/or Diastolic blood pressure more than or equal to 100 mmHg)
* If taking more than or equal to 2 blood pressure medications at the time of screening
* Systolic blood pressure more than 180 and/or Diastolic blood pressure more than or equal to 120 mmHg at any point in the study
* Present or past history of major cardiovascular disease including myocardial infarction, angina, cardiac arrhythmia, heart failure, stroke, transient ischemic attack, or seizure.
* Pregnant or breastfeeding individuals
* History of kidney disease
* History of insulin requiring diabetes
* Estimated glomerular filtration rate less than 60ml/min/1.73 m2, albumin creatinine ratio more than or equal to 30 mg/g
* Hepatic transaminase levels more than 3 times the upper limit of normal
* Anemia (men, Hb less than 13 g/dL; women, Hb less than 12 g/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in 24h mean Systolic Blood Pressure (SBP) | 3 weeks
  Difference in the change in 24h mean SBP following high and low salt diets, between the polygenic score groups.
Change in N-terminal pro-B-type Natriuretic Peptide (NTproBNP) (NTproBNP) | 3 weeks
  Difference in the change in NTproBNP levels following high and low salt diets, between the the polygenic score groups.

SECONDARY OUTCOMES:
Change in 24h mean Diastolic Blood Pressure (DBP) | 3 weeks
  Difference in the change in the 24h mean DBP following high and low salt diets between the polygenic score groups.
Change in Daytime Diastolic Blood Pressure (DBP) | 3 weeks
  Difference in the change in the Daytime DBP following high and low salt diets between the polygenic score groups.
Change in Nighttime Diastolic Blood Pressure (DBP) | 3 weeks
  Difference in the change in the Nighttime DBP following high and low salt diets between the polygenic score groups.
Change in Daytime Systolic Blood Pressure (SBP) | 3 weeks
  Difference in the change in the Daytime SBP following high and low salt diets between the polygenic score groups.
Change in Nighttime Systolic Blood Pressure (SBP) | 3 weeks
  Difference in the change in the Nighttime SBP following high and low salt diets between the polygenic score groups.
Change in 24h Urinary Excretion (Sodium) | 3 weeks
  Difference in the change in 24h urinary excretion (sodium) following high and low salt diets between the polygenic score groups.
Change in 24h Urinary Excretion (Potassium) | 3 weeks
  Difference in the change in 24h urinary excretion (potassium) following high and low salt diets between the polygenic score groups.
Change in Daytime Urinary Excretion (Sodium) | 3 weeks
  Difference in the change Daytime urinary excretion (sodium) following high and low salt diets between the polygenic score groups.
Change in Daytime Urinary Excretion (Potassium) | 3 weeks
  Difference in the change in Daytime urinary excretion (potassium) following high and low salt diets between the polygenic score groups.
Change in Nighttime Urinary Excretion (Sodium) | 3 weeks
  Difference in the change in Nighttime urinary excretion (sodium) following high and low salt diets between the polygenic score groups.
Change in Nighttime Urinary Excretion (Potassium) | 3 weeks
  Difference in the change in Nighttime urinary excretion (potassium) following high and low salt diets between the polygenic score groups.
Change in Natriuretic Peptide Levels (BNP) | 3 weeks
  Difference in the change in BNP levels following high and low salt diets between the polygenic score groups
Change in Natriuretic Peptide Levels (MRproANP) | 3 weeks
  Difference in the change in MRproANP levels following high and low salt diets between the polygenic score groups
Change in Natriuretic Peptide Levels (BNP) with Volume Loading | 3 weeks
  Difference in the change in BNP with the volume loading protocol (from start to end of protocol) after high and low salt diets between the genotype groups.
Change in Natriuretic Peptide Levels (NTproBNP) with Volume Loading | 3 weeks
  Difference in the change in NTproBNP with the volume loading protocol (from start to end of protocol) after high and low salt diets between the genotype groups.
Change in Natriuretic Peptide Levels (MRproANP) with Volume Loading | 3 weeks
  Difference in the change in MRproANP with the volume loading protocol (from start to end of protocol) after high and low salt diets between the genotype groups.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, FAHA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided